CLINICAL TRIAL: NCT06676813
Title: Effect of Alternate Day Fasting Over Standard Medical Management Alone to Reverse Non-alcoholic Steatohepatitis(NASH), A Randomized Controlled Trial. FAST Trial"
Brief Title: Effect of Alternate Day Fasting Over Standard Medical Management Alone to Reverse Non-alcoholic Steatohepatitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/8/2023-ACAD/E-12745/680
Record Dates: First submitted 2024-06-22; First posted 2024-11-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-06

CONDITIONS: Non Alcoholic Steatohepatitis
Keywords: Alternate day fasting.; NASH; MASH; Steatotic liver disease; Cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADF (Experimental): Experimental: Alternate day fasting, along with standard medical management.
  Interventions: Behavioral: Alternate day fasting
- Control arm (No Intervention): Standard medical management.

INTERVENTIONS:
Behavioral: Alternate day fasting — Alternate day fasting
  Arms: ADF

SUMMARY:
The aims of this study are as follows: To compare the role of alternate-day fasting over standard medical management alone to reverse NASH.

DETAILED DESCRIPTION:
Emerging evidence suggests the role of alternate-day fasting (ADF) in patients with obesity and fatty liver. It helps to lose weight and improvement in liver fat content. ADF regimen protocol includes fast day(restricted calorie intake and time-specific feeding) and feast day(ad libitum feed over 24 hours). Lowering the weight and improvement of the fatty liver. NASH is a prevalent cause of liver disease. Literature is evident that ADF improves fatty liver and metabolic components, and NASH improves with weight loss. Still, data about the role of ADF in the management of NASH is lacking. Hence, this study focuses on the role of ADF in NASH.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years. BMI 25-40kg/m3, and CAP more than 290
* Stable weight in the last 3 months prior to enrolling in the study(<5kg weight variation)
* Imaging showed steatotic liver disease, liver stiffness <14kPa measured by fibroscan
* Histologically proven NASH/MASH, fibrosis up to F3
* Subjects willing to participate in the study

Exclusion Criter

* Liver stiffness >14kPa measured by fibroscan or Fibrosis >F3
* Diabetes with HbA1c>8.5%
* Patients with another co-existing active liver disease e.g. hepatitis B or C, alcoholic liver disease
* Patients with cirrhosis, hepatocellular carcinoma(HCC), or other malignancy
* Chronic kidney disease, cardiovascular disorders, uncontrolled hypertension
* Chronic infections, chronic inflammatory diseases
* Patients on weight loss medications e.g semaglutide
* Pregnant or lactating women and those planning a pregnancy A patient who is not willing to participate in the study or failed to provide the consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of NASH over a 24-week duration. | 24 weeks
  Histologically confirmed NASH, biochemical resolution.

SECONDARY OUTCOMES:
Change in the quality of life index | Change from baseline to 24 weeks
  The investigators will assess the CLDQ-NASH score (Chronic Liver Disease Questionnaire for Nonalcoholic Steatohepatitis), which comprises 29 items rated on a scale from 1 to 7. Each item score reflects the patient's experience, with 1 indicating the worst and 7 indicating the best quality of life.
  The average score across all 29 items provides an overall quality of life result:
  * 1 to 3: Indicates a poor quality of life, with significant symptom burden and substantial impact on daily activities.
  * 4 to 5: Suggests a moderate quality of life, where symptoms are present but manageable, with some limitations in daily activities.
  * 6 to 7: Reflects a high quality of life, with minimal symptoms and few or no limitations on daily life.
Change in stage of fibrosis | Change from baseline to 24 weeks
  Measured by fibroscan(LSM)
Weight | Change from baseline to 24 weeks
  Change in weight at 1, 3, and 6 month of follow up.
Change in glycaemic status | Change from baseline to 24 weeks
  Change in HbA1c level at baseline, 3 and 6 months.
Change in liver fat content | Change from baseline to 24 weeks
  Measured by fibroscan(CAP)
Change in bone mineral density | Change from baseline to 24 weeks
  As measured by dual-energy X ray absorptiometry (DEXA) scan
Change in faecal microbiota. | Change from baseline to 24 weeks
  Stool analysis
Body mass index | 24 weeks
  Change in body mass index at 1, 3, and 6 month of follow up.
Waist to hip ratio | 24 weeks
  Change in Waist to hip ratio at 1, 3, and 6 month of follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, Delhi, India

IPD SHARING:
Plan to Share IPD: No
Investigators currently do not plan to share individual participant data (IPD) from this study. The decision is based on considerations of patient privacy, confidentiality concerns, and the lack of a data-sharing infrastructure. While the aggregated study results will be published and made publicly available, sharing individual-level data could pose risks related to identifying participants. Therefore, IPD will not be shared beyond what is required for regulatory purposes.

REFERENCES:
- [Background] Teng ML, Ng CH, Huang DQ, Chan KE, Tan DJ, Lim WH, Yang JD, Tan E, Muthiah MD. Global incidence and prevalence of nonalcoholic fatty liver disease. Clin Mol Hepatol. 2023 Feb;29(Suppl):S32-S42. doi: 10.3350/cmh.2022.0365. Epub 2022 Dec 14. PMID 36517002
- [Background] Carr RM, Oranu A, Khungar V. Nonalcoholic Fatty Liver Disease: Pathophysiology and Management. Gastroenterol Clin North Am. 2016 Dec;45(4):639-652. doi: 10.1016/j.gtc.2016.07.003. Epub 2016 Oct 13. PMID 27837778
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ. The diagnosis and management of non-alcoholic fatty liver disease: practice Guideline by the American Association for the Study of Liver Diseases, American College of Gastroenterology, and the American Gastroenterological Association. Hepatology. 2012 Jun;55(6):2005-23. doi: 10.1002/hep.25762. No abstract available. PMID 22488764
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Castro Narro GE, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. Hepatology. 2023 Dec 1;78(6):1966-1986. doi: 10.1097/HEP.0000000000000520. Epub 2023 Jun 24. PMID 37363821
- [Background] Loomba R, Wong R, Fraysse J, Shreay S, Li S, Harrison S, Gordon SC. Nonalcoholic fatty liver disease progression rates to cirrhosis and progression of cirrhosis to decompensation and mortality: a real world analysis of Medicare data. Aliment Pharmacol Ther. 2020 Jun;51(11):1149-1159. doi: 10.1111/apt.15679. Epub 2020 May 5. PMID 32372515
- [Background] Rinella ME, Neuschwander-Tetri BA, Siddiqui MS, Abdelmalek MF, Caldwell S, Barb D, Kleiner DE, Loomba R. AASLD Practice Guidance on the clinical assessment and management of nonalcoholic fatty liver disease. Hepatology. 2023 May 1;77(5):1797-1835. doi: 10.1097/HEP.0000000000000323. Epub 2023 Mar 17. No abstract available. PMID 36727674
- [Background] Sanyal AJ, Chalasani N, Kowdley KV, McCullough A, Diehl AM, Bass NM, Neuschwander-Tetri BA, Lavine JE, Tonascia J, Unalp A, Van Natta M, Clark J, Brunt EM, Kleiner DE, Hoofnagle JH, Robuck PR; NASH CRN. Pioglitazone, vitamin E, or placebo for nonalcoholic steatohepatitis. N Engl J Med. 2010 May 6;362(18):1675-85. doi: 10.1056/NEJMoa0907929. Epub 2010 Apr 28. PMID 20427778
- [Background] Promrat K, Kleiner DE, Niemeier HM, Jackvony E, Kearns M, Wands JR, Fava JL, Wing RR. Randomized controlled trial testing the effects of weight loss on nonalcoholic steatohepatitis. Hepatology. 2010 Jan;51(1):121-9. doi: 10.1002/hep.23276. PMID 19827166
- [Background] van den Hoek AM, de Jong JCBC, Worms N, van Nieuwkoop A, Voskuilen M, Menke AL, Lek S, Caspers MPM, Verschuren L, Kleemann R. Diet and exercise reduce pre-existing NASH and fibrosis and have additional beneficial effects on the vasculature, adipose tissue and skeletal muscle via organ-crosstalk. Metabolism. 2021 Nov;124:154873. doi: 10.1016/j.metabol.2021.154873. Epub 2021 Sep 1. PMID 34478753
- [Background] Sullivan S, Kirk EP, Mittendorfer B, Patterson BW, Klein S. Randomized trial of exercise effect on intrahepatic triglyceride content and lipid kinetics in nonalcoholic fatty liver disease. Hepatology. 2012 Jun;55(6):1738-45. doi: 10.1002/hep.25548. Epub 2012 Apr 25. PMID 22213436
- [Background] Yang W, Cao M, Mao X, Wei X, Li X, Chen G, Zhang J, Wang Z, Shi J, Huang H, Yao X, Liu C. Alternate-day fasting protects the livers of mice against high-fat diet-induced inflammation associated with the suppression of Toll-like receptor 4/nuclear factor kappaB signaling. Nutr Res. 2016 Jun;36(6):586-93. doi: 10.1016/j.nutres.2016.02.001. Epub 2016 Feb 16. PMID 27188904
- [Background] Wei X, Lin B, Huang Y, Yang S, Huang C, Shi L, Liu D, Zhang P, Lin J, Xu B, Guo D, Li C, He H, Liu S, Xue Y, Xu Y, Zhang H. Effects of Time-Restricted Eating on Nonalcoholic Fatty Liver Disease: The TREATY-FLD Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e233513. doi: 10.1001/jamanetworkopen.2023.3513. PMID 36930148
- [Background] Cai H, Qin YL, Shi ZY, Chen JH, Zeng MJ, Zhou W, Chen RQ, Chen ZY. Effects of alternate-day fasting on body weight and dyslipidaemia in patients with non-alcoholic fatty liver disease: a randomised controlled trial. BMC Gastroenterol. 2019 Dec 18;19(1):219. doi: 10.1186/s12876-019-1132-8. PMID 31852444
- [Background] Hatori M, Vollmers C, Zarrinpar A, DiTacchio L, Bushong EA, Gill S, Leblanc M, Chaix A, Joens M, Fitzpatrick JA, Ellisman MH, Panda S. Time-restricted feeding without reducing caloric intake prevents metabolic diseases in mice fed a high-fat diet. Cell Metab. 2012 Jun 6;15(6):848-60. doi: 10.1016/j.cmet.2012.04.019. Epub 2012 May 17. PMID 22608008